CLINICAL TRIAL: NCT04822636
Title: Family Mental Health Family Navigator
Brief Title: Family Mental Health Family Navigator Project (FMHN)
Acronym: FMHN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: San Francisco General Hospital Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1929675
Record Dates: First submitted 2021-03-25; First posted 2021-03-30 (Actual); Last update posted 2025-04-07 (Actual); Status verified 2025-04

CONDITIONS: Mental Health
Keywords: Adolescent; Publicly-insured Youth; Mental Health; Navigator Service; Access; Children
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: This is a within-person, pre-post design in which the investigators will test a theory-driven, family-based navigator treatment engagement intervention (FMHN) while also collecting data on the FMHN model's potential implementation and adoption within a public hospital and behavioral health settings.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Family-based mental health navigation (Experimental): Family-based navigator intervention combined with mHealth practices to improve mental health treatment initiation and engagement
  Interventions: Behavioral: Family-based mental health navigation

INTERVENTIONS:
Behavioral: Family-based mental health navigation — Family-based navigator intervention combined with mHealth practices to improve mental health treatment initiation and engagement

SUMMARY:
This study will focus on developing and testing a family-based mental health navigator intervention, the Family Mental Health Navigator (FMHN), to evaluate whether the intervention combined with mHealth is preliminary efficacious in improving mental health service initiation and engagement for publicly-insured youth.

DETAILED DESCRIPTION:
The study will demonstrate how a family-based navigator intervention combined with mHealth may lead to improved mental health treatment initiation and engagement among publicly-insured youth. Publicly-insured youth have high rates of mental health symptoms relative to youth in the community, and are disproportionately racial and ethnic minorities, only perpetuating disparities in this population's mental health access and engagement. The proposed project will develop and test a family-based navigator intervention, the Family Mental Health Navigator (FMHN), a natural fit for improving publicly-insured youth's mental health service and clinical outcomes. The study will start with identifying the feasibility and acceptability of the FMHN intervention. Then, the study will determine whether the FMHN intervention improves publicly-insured youth mental health treatment initiation and engagement. Finally, the study will characterize patterns of pre- and post-service outcomes along the behavioral health services cascade of care, to further evaluate the feasibility, acceptability, and preliminary impact of the FMHN model.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking and/or Spanish-speaking youth
* Ages 6-17
* Are currently receiving services at the San Francisco General Hospital
* Are publicly insured
* Have an involved caregiver/legal guardian for consent
* Family has mobile phone access

Exclusion Criteria:

* Youth is not English-speaking nor Spanish-speaking
* Caregiver has impairment that would preclude providing informed consent
* Unavailable guardian for consent

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2022-06-06 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Time to treatment referral | 12 months post enrollment
  Number of days until treatment referral is made
Time to treatment initiation | 12 months post enrollment
  Number of days until attendance at first treatment session
Treatment engagement | 12 months post enrollment
  Engagement as measured by attendance in treatment for 6 or more weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marina Tolou-Shams, Ph.D, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Zuckerberg San Francisco General Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No